CLINICAL TRIAL: NCT03304392
Title: Advancing Mental Health Care by Improving the Delivery of Therapist-guided, Internet-delivered Cognitive Behavioural Therapy in Clinical Practice
Brief Title: Therapist-guided Internet-delivered Cognitive Behavioural Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 375860
Record Dates: First submitted 2017-09-29; First posted 2017-10-09 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-11

CONDITIONS: Anxiety; Depression
Keywords: anxiety; depression; internet-delivered cognitive behaviour therapy; randomized controlled trial; patient-centered; knowledge implementation; mental health system; therapist-assistance
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized ICBT (Experimental): An 8-week transdiagnostic internet-delivered cognitive behavioural therapy (ICBT) will be delivered to participants. All clients will receive support from registered social workers, psychologists or supervised graduate students, with experience delivering ICBT, with contact depending upon group allocation. In addition to the online program, therapists, registered social workers, psychologists or supervised graduate students, with experience delivering ICBT will provide support within one business day of client emails. Amount of contact will be personalized to patients' needs.
  Interventions: Behavioral: Personalized ICBT
- Standard ICBT (Active Comparator): An 8-week transdiagnostic internet-delivered cognitive behavioural therapy (ICBT) will be delivered to participants. All clients will receive support from registered social workers, psychologists or supervised graduate students, with experience delivering ICBT, with contact depending upon group allocation. In addition to the online program, therapists, registered social workers, psychologists or supervised graduate students, with experience delivering ICBT will provide support by email only once a week. Therapist will spend approximately 15 minutes per week/per client.
  Interventions: Behavioral: Standard ICBT

INTERVENTIONS:
Behavioral: Personalized ICBT — An 8-week transdiagnostic internet-delivered cognitive behavioural therapy (ICBT) will be delivered to participants. All clients will receive support from registered social workers, psychologists or supervised graduate students, with experience delivering ICBT, with contact depending upon group allocation. In addition to the online program, therapists, registered social workers, psychologists or supervised graduate students, with experience delivering ICBT will provide support within one business day of client emails. Amount of contact will be personalized to patients' needs.
  Arms: Personalized ICBT
Behavioral: Standard ICBT — An 8-week transdiagnostic internet-delivered cognitive behavioural therapy (ICBT) will be delivered to participants. All clients will receive support from registered social workers, psychologists or supervised graduate students, with experience delivering ICBT, with contact depending upon group allocation. In addition to the online program, therapists, registered social workers, psychologists or supervised graduate students, with experience delivering ICBT will provide support by email only once a week. Therapist will spend approximately 15 minutes per week/per client.
  Arms: Standard ICBT

SUMMARY:
Depression and anxiety are prevalent and disabling conditions that often go untreated. Internet-delivered Cognitive Behaviour Therapy (ICBT) is a relatively new approach to treatment that is a convenient way for patients to access care. ICBT is typically highly standardized and involves patients reviewing weekly lessons over the Internet. Patients also receive brief weekly support from a therapist via secure emails or phone calls. Past research shows that ~75% of patients complete ICBT and report large symptom improvements. Although these results are very promising, research also suggests that ICBT could potentially be improved by being more personalized in terms of amount of therapist contact, especially for clients with more severe symptoms. The current trial will involve therapists who work in a clinic that specializes in ICBT. Over one year, 440 patients with depression and/or anxiety will be randomized to either receive standardized (5 lessons completed in 8 weeks; once week therapist contact) or personalized ICBT (5 lessons completed in 8 weeks; personalized therapist contact depending on needs of patient). Psychosocial outcomes of patients in the two treatment arms will be compared post-treatment and at 3-month, 6-month, and 1-year follow-up from enrollment. Data on intervention usage, satisfaction measures, and costs will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* residing in Saskatchewan, Canada
* endorsing symptoms of anxiety or depression
* able to access a computer and internet service
* willing to provide a physician as emergency contact

Exclusion Criteria:

* high suicide risk
* suicide attempt or hospitalization in the last year
* primary problems with psychosis, alcohol or drug problems, mania
* currently receiving active psychological treatment for anxiety or depression
* not present in province during treatment; concerns about online therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Change in depression | baseline, start of each Lesson 2-5, 8 weeks, 3 months, 6 months, and 1 year follow up
  Measured by Patient Health Questionnaire - 9 Item (PHQ-9)
Change in anxiety | baseline, start of each Lesson 2-5, 8 weeks, 3 months, 6 months, and 1 year follow up
  Measured by Generalize Anxiety Disorder - 7 Item (GAD7)

SECONDARY OUTCOMES:
Change in psychological distress | baseline, 8 weeks, 3 months, 6 months, and 1 year follow up
  Measured by Kessler 10-Item Scale
Change in disability | baseline, 8 weeks, 3 months, 6 months, and 1 year follow up
  Measure by Sheehan Disability Scale-3 Item
Change in panic symptoms | baseline, 8 weeks, 3 months, 6 months, and 1 year follow up
  Measured by Panic Disorder Severity Scale-Self Report
Change in social anxiety symptoms | baseline, 8 weeks, 3 months, 6 months, and 1 year follow up
  Measured by Social Interaction Anxiety Scale
Change in social phobia symptoms | baseline, 8 weeks, 3 months, 6 months, and 1 year follow up
  Measured by Social Phobia Scale-Short form
Change in post-traumatic symptoms | Administered to only those participants meeting criteria for post-traumatic stress based on the modified brief Life Events Checklist for DSM 5 (LEC-5) at each time point: baseline, 3 months, 6 months, and 1 year follow up
  Measured by PTSD Checklist 5
Change in quality of life symptoms | baseline, 8 weeks, 3 months, 6 months, and 1 year follow up
  Measured by EQ-5D-5L
Change in treatment costs | Part 1 and 2: baseline, 3 months, 6 months, and 1 year follow up; Part 3: baseline and 1 year follow up
  Measured by Treatment Inventory of Costs in Psychiatric Patients (TIC-P) Adapted for Canada
Therapeutic alliance | 8 weeks
  Measured by Working Alliance Inventory-Short Form
Treatment credibility | baseline and 8 weeks
  Measured by Credibility Questionnaire
Treatment satisfaction | 8 weeks
  Measured by Internet-CBT Treatment Satisfaction Measure
Engagement | 8 weeks
  Measured by: number of lessons completed, number of days of access, number of emails sent to therapist, number of phone calls with therapist, number of emails from therapist to client, total words emailed to therapist, total words emailed from therapist to patient

CONTACTS AND LOCATIONS:
Overall Officials: Heather D Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- Online Therapy Unit, University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No